CLINICAL TRIAL: NCT00372463
Title: Internet Diabetes Self-Management: A Randomized Trial
Brief Title: Internet Diabetes Self-Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 49148
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; type 2 diabetes; type II diabetes; diabetes mellitus; diabetes type 2; diabetes type II; diabetes education; patient education; workshop; class; education; online; on-line; internet; web
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Behavioral: 6-week Online Diabetes Self-Management Educational Program

SUMMARY:
Diabetes is a growing health problem causing personal suffering, comorbid conditions, premature death, and high costs to the individual, the health care system and society. Many of these problems can be prevented or delayed by controlling the disease. This in turn requires daily self-management by patients.

We will evaluate an Internet based small group Diabetes Self-Management Program. This program will be adapted from the Chronic Disease Self-Management Program Online, already developed and currently being evaluated by the investigators. Participants with type 2 diabetes will be randomized to participate in the Internet Program or serve as controls continuing with usual care. Treatment subjects will participate in a structured 6 week interactive web-based online class with 20-24 other participants and 2 trained peer moderators.

If successful, this project will result in a new and effective means of reaching the CDC objective and more importantly in improving the quality of life and health status of people with diabetes while reducing health care utilization and thus costs.

DETAILED DESCRIPTION:
Diabetes is a growing health problem causing personal suffering, comorbid conditions, premature death, and high costs to the individual, the health care system and society. Many of these problems can be prevented or delayed by controlling the disease. This in turn requires daily self-management by patients.

The CDC has recognized the importance of self-management by setting a 2010 objective of having 60% of diabetics receive diabetes education. Unfortunately, many people cannot receive such education because it is not available or they do not wish to or cannot participate in small group or one on one education.

The Internet may offer a viable alternative. We will evaluate an Internet based small group Diabetes Self-Management Program. This program will be adapted from the Chronic Disease Self-Management Program Online, already developed and currently being evaluated by the investigators. Participants with type 2 diabetes will be randomized to participate in the Internet Program or serve as controls continuing with usual care. Treatment subjects will participate in a structured 6 week interactive web-based online class with 20-24 other participants and 2 trained peer moderators.

Data will be collected online at baseline, 6 months and 1 year. Outcome measures include health related quality of life (fatigue, physical discomfort, the symptoms of hypoglycemia and hyperglycemia, activity limitations, health distress, and self-rated health), metabolic control (hemoglobin A1c), health care utilization (decreases in outpatient visits to physicians, increases in the percentage of participants having received an eye examination in the past year, increases in the number of times a health professional has examined participants' feet, and decreases in emergency department visits, hospitalizations, and hospital days), health behaviors (aerobic exercise, communication with physicians, diet, glucose self-monitoring, and self-examination of the feet), and self-efficacy to manage diabetes.

If successful, this project will result in a new and effective means of reaching the CDC objective and more importantly in improving the quality of life and health status of people with diabetes while reducing health care utilization and thus costs.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Live in the United States
* Access to internet and an email account

Exclusion Criteria:

* Under 18 years of age
* Pregnant
* Treatment for cancer in past 12 months
* Have taken any Stanford self-management program previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2006-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Health related-quality of life
Metabolic control (HbA1c)
Heath care utilization
Behaviors
Self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lorig, DrPH, Principal Investigator — Stanford University; Diana Laurent, MPH, Study Director — Stanford University
Locations (1):
- Stanford Patient Education Research Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Case S, Jernigan V, Gardner A, Ritter P, Heaney CA, Lorig KR. Content and frequency of writing on diabetes bulletin boards: does race make a difference? J Med Internet Res. 2009 Jun 24;11(2):e22. doi: 10.2196/jmir.1153. PMID 19632975